CLINICAL TRIAL: NCT01277588
Title: Evaluation of the Physicians and Patients Experience of Fetal Scalp Sampling
Status: Completed | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Maria Jonsson, M.D., Ph.D. Consultant, Uppsala University Hospital
Other Study IDs: UAS2010/003
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Questionnaire; Fetal Scalp Sampling
Keywords: fetal scalp sampling; experience questionnaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient
- Physcician

SUMMARY:
During labor, fetal scalp sampling is performed if the CTG registration is abnormal. The test is performed with the woman in the supine position and is generally described as a difficult and cumbersome procedure.

DETAILED DESCRIPTION:
Women who were subjected to fetal scalp sampling are asked to fill in a questionnaire within 24 hours after delivery. The questionnaire deals with how the woman experienced the testing procedure.

Physicans who performed the test are asked to fill in a questionnaire within 24 hours after delivery. The questionnaire deals with how the physician experienced the testing procedure.

ELIGIBILITY:
Inclusion Criteria:

* fetal scalp sampling during labor

Exclusion Criteria:

* non-proficiency in the Swedish language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who are subjected to fetal scalp sampling during labor Physicians performning fetal scalp sampling
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of obstetrics and gynecology, Uppsala, Sweden